CLINICAL TRIAL: NCT01685476
Title: Validation of a New Non Invasive Method for Intracranial Pressure Monitoring
Brief Title: NIMI-NICU: Non Invasive Monitoring of the Intracranial Pressure - NeuroIntensive Care Unit
Acronym: MINIPIC REA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Echodia SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: CHU-0124; 2010-A00509-30
Record Dates: First submitted 2012-08-31; First posted 2012-09-14 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Intracranial Pressure; Traumatic Brain Injury; Stroke; Intracranial Hemorrhages
Keywords: Cochlear microphonic potential; non invasive method; indirect monitoring; intracranial pressure
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke; Intracranial Hemorrhages

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Intracranial pressure (Other)
  Interventions: Device: Echodia® hand-held equipment

INTERVENTIONS:
Device: Echodia® hand-held equipment

SUMMARY:
In clinical practice, intracranial pressure (ICP) represents a key parameter for diagnosing and treating several conditions. Physicians having to manage cases of head trauma, stroke and hydrocephalus need to assess the time course of ICP, yet they are often unwilling to implement invasive monitoring beyond the acute stage, on account of high septic risks. Standard techniques include direct ventricular manometry or measurement in the parenchyma with electronic or fiberoptic devices. Therefore, the design of non-invasive clinical methods for gaining access to pressure changes is an important challenge. Fluctuations of ICP are transmitted to the fluid spaces of the inner ear through the cochlear aqueduct. The Biophysics Laboratory (School of Medicine of Clermont-Ferrand) described that the intra-labyrinthic pressure modify the functional activities of the outer hair cells in the cochlea. Thereby, increases in ICP are transferred to increases in intra-cochlear pressure, which is detected as modifications in cochlear activities. Cochlear activities' recording are non-invasive and technically simple. A probe is gently inserted into the outer portion of the external ear canal.

The objective of this study is to assess prospectively the accuracy and the precision of a new method for ICP monitoring (using cochlear activities) compared with invasive gold standard CSF pressure monitoring.

DETAILED DESCRIPTION:
The purpose of this study is to examine the evolution of the electrophysiological cochlear activity (cochlear microphonic potential, CMP), with a non invasive method, during invasive ICP monitoring. The data analysis will determine relationship between ICP variations and CMP variations.

Continuous ICP monitoring has an important place in neuro-intensive care. ICP may be measured either within the ventricular cerebrospinal fluid or within the brain parenchyma.

The purpose of this study is to assess prospectively the accuracy and the precision of a new method for indirect ICP monitoring (using electrophysiological cochlear activity) compared with an invasive gold standard ICP monitoring. The data analysis will determine relationship between ICP variations and CMP variations.

Electrophysiological cochlear activities, so called electrocochleography (ECochG), are a non invasive and totally passive method used in routine in ENT department. The response measured in ECochG is the cochlear microphonic potential (CMP), generated by the outer hair cells following by presenting tone burst at 1kHz. CMP is recorded with the help of an Echodia® hand-held equipment.

Technically, a simple, non-invasive detection of ICP changes and ICP monitoring can be afforded by CMP recordings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intracranial pressure monitoring
* Age greater than 18
* consent form signed by a close relative (husband, wife, children, legal guardian),
* Patient covered under French social security or being a beneficiary of such a regime under the terms of the Act of August 9, 2004

Exclusion Criteria:

* Refusal by the close relative to sign a consent form
* Impossibility of electrophysiological measurements (pathophysiological reason)
* Technical troubles with the device
* Patient uncovered under French social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Cochlear Microphonic Potential phase shift | acquisition every 5minutes during 4hours

SECONDARY OUTCOMES:
IntraCranialPressure variations | every minutes during 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Laurent SAKKA, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Giraudet F, Longeras F, Mulliez A, Thalamy A, Pereira B, Avan P, Sakka L. Noninvasive detection of alarming intracranial pressure changes by auditory monitoring in early management of brain injury: a prospective invasive versus noninvasive study. Crit Care. 2017 Feb 21;21(1):35. doi: 10.1186/s13054-017-1616-2. PMID 28219399